CLINICAL TRIAL: NCT01241292
Title: Phase 1 Multiple Ascending Dose Study of Elotuzumab (BMS-901608) in Combination With Lenalidomide/Low-dose Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma in Japan
Brief Title: Japanese Study of BMS-901608 (Elotuzumab) in Combination With Lenalidomide and Low Dose Dexamethasone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA204-005
Record Dates: First submitted 2010-11-04; First posted 2010-11-16 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BMS-901608 (Elotuzumab) 10mg (Experimental)
  Interventions: Biological: BMS-901608 (Elotuzumab) 10 mg
- BMS-901608 (Elotuzumab) 20mg (Experimental)
  Interventions: Biological: BMS-901608 (Elotuzumab) 20 mg

INTERVENTIONS:
Biological: BMS-901608 (Elotuzumab) 10 mg — Injection, Intravenous, 10 mg/kg, Weekly at cycle 1 and 2, bi-weekly at cycle 3 and thereafter, Until disease progression or unacceptable toxicity became apparent
  Arms: BMS-901608 (Elotuzumab) 10mg
Biological: BMS-901608 (Elotuzumab) 20 mg — Injection, Intravenous, 20 mg/kg, Weekly at cycle 1 and 2, bi-weekly at cycle 3 and thereafter, Until disease progression or unacceptable toxicity became apparent
  Arms: BMS-901608 (Elotuzumab) 20mg

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Elotuzumab when given in combination with Lenalidomide and low-dose Dexamethasone in subjects with relapsed or refractory multiple myeloma (MM) in Japan.

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Received between 1 to 4 prior lines of therapy
* Measureable disease
* Men and women of childbearing potential (WOCBP) must be using two acceptable methods of contraception
* Men must agree to use a latex condom and a second form of birth control during sexual contact with WOCBP and must agree to not donate semen during study drug therapy
* Subjects must be willing to refrain from blood donations during study drug therapy

Exclusion Criteria:

* Subjects with non-secretory or oligo-secretory or light-chain only myeloma or active/prior plasma cell leukemia or known /suspect POEMS syndrome
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
* Unable to take aspirin daily as prophylactic anticoagulation therapy. Prior history of inability to tolerate weekly 40 mg dexamethasone
* History of renal failure
* History of clinical significant thrombosis, such as treatment for thrombosis was required

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2017-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Niigata, Niigata

REFERENCES:
- [Derived] Iida S, Nagai H, Kinoshita G, Miyoshi M, Robbins M, Pandya D, Bleickardt E, Chou T. Elotuzumab with lenalidomide and dexamethasone for Japanese patients with relapsed/refractory multiple myeloma: phase 1 study. Int J Hematol. 2017 Mar;105(3):326-334. doi: 10.1007/s12185-016-2138-4. Epub 2016 Nov 15. PMID 27848182
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seven participants were enrolled and 6 entered the treatment period. Reason for 1 participant not entering treatment period: participant no longer met study criteria.
Groups:
- Elotuzumab 10 mg/kg: Elotuzumab 10 mg/kg was intravenously (IV) given weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity. Elotuzumab was first given at 10 mg/kg. If all participants completed the first cycle and none experienced a dose limiting toxicity (DLT), the dose was escalated to 20 mg/kg. If 1 experienced a DLT at 10 mg/kg, 3 additional participants were assigned to 10 mg/kg. If no additional participants experienced a DLT, the dose was escalated to 20 mg/kg. Lenalidomide 25 mg was administered orally once daily for the first 3 weeks of each 4-week cycle. On weeks without elotuzumab, dexamethasone was administered as a single oral (PO) dose of 40 mg. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (3 to 24 hours prior to the start of elotuzumab) and 8 mg IV (45 min prior to start of elotuzumab).
- Elotuzumab 20 mg/kg: Elotuzumab 20 mg/kg was intravenously (IV) given weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity. Elotuzumab was first given at 10 mg/kg. If all participants completed the first cycle and none experienced a dose limiting toxicity (DLT), the dose was escalated to 20 mg/kg. If 1 experienced a DLT at 10 mg/kg, 3 additional participants were assigned to 10 mg/kg. If no additional participants experienced a DLT, the dose was escalated to 20 mg/kg. Lenalidomide 25 mg was administered orally once daily for the first 3 weeks of each 4-week cycle. On weeks without elotuzumab, dexamethasone was administered as a single oral (PO) dose of 40 mg. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (3 to 24 hours prior to the start of elotuzumab) and 8 mg IV (45 min prior to start of elotuzumab).
Period: Overall Study
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Started | 3 | 3
Entered Treatment Period | 3 | 3
Completed | 0 (completed=treatment on-going) | 0 (completed=treatment on-going)
Not Completed | 3 | 3
Not completed — Administrative Reason by Sponsor | 1 | 0
Not completed — Disease Progression | 2 | 0
Not completed — Study Drug Toxicity | 0 | 1
Not completed — Participant Discontinued Treatment | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug were summarized.
Groups:
- Elotuzumab 10 mg/kg: Elotuzumab was intravenously (IV) injected at a dose of 10 mg/kg weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity became apparent. Lenalidomide 25 mg was administered orally once daily for the first 3 weeks of each 4-week cycle. The dose of lenalidomide was administered at least 2-4 hours after completion of elotuzumab infusion. On weeks without elotuzumab administration, dexamethasone was administered as a single dose of 40 mg PO. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (between 3 to 24 hours prior to the start of the elotuzumab infusion) and 8 mg IV (At least 45 min prior to the start of the elotuzumab infusion).
- Elotuzumab 20 mg/kg: Elotuzumab was intravenously (IV) injected at a dose of 20 mg/kg weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity became apparent. Lenalidomide 25 mg was administered orally once daily for the first 3 weeks of each 4-week cycle. The dose of lenalidomide was administered at least 2-4 hours after completion of elotuzumab infusion. On weeks without elotuzumab administration, dexamethasone was administered as a single dose of 40 mg PO. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (between 3 to 24 hours prior to the start of the elotuzumab infusion) and 8 mg IV (At least 45 min prior to the start of the elotuzumab infusion).
- Total: Total of all reporting groups
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 61.0 [52 to 66] | 66.0 [60 to 75] | 63.5 [52 to 75]
Age, Customized [Number; unit: participants]
  Less than (<) 65 | 2 | 1 | 3
  65 to < 75 | 1 | 1 | 2
  Greater than, equal to 75 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, Deaths
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4= Potentially Life-threatening or disabling. Data cut-off February 2014.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized (Treated Participants).
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants
  All SAEs Any Grade | 2 | 3
  Grade 3-4 SAEs | 1 | 3
  AEs Leading to Discontinuation | 0 | 1
  Grade 3-4 AEs | 3 | 3
  Deaths | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Relevant Vital Sign Findings
Description: Vital signs (body temperature, seated blood pressure, heart rate, and respiration rate) were recorded at screening on Days 1, 8, 15, and 22 of Cycles 1 and 2, on Days 1 and 15 of Cycle 3, and at the end of treatment. Blood pressure (Diastolic and Systolic) and heart rate were recorded after the participant sat quietly for at least 5 minutes. Clinical relevance of vital sign data was determined by the investigator.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized.
Measure: Number; unit: participants
Groups:
- Elotuzumab 10 mg/kg: Elotuzumab was administered IV at a dose of 10 mg/kg weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity became apparent. Lenalidomide 25 mg was administered PO once daily for the first 3 weeks of each 4-week cycle. The dose of lenalidomide was administered at least 2-4 hours after completion of elotuzumab infusion. On weeks without elotuzumab administration, dexamethasone was administered PO as a single dose of 40 mg. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (between 3 to 24 hours prior to the start of the elotuzumab infusion) and 8 mg IV (At least 45 min prior to the start of the elotuzumab infusion).
- Elotuzumab 20 mg/kg: Elotuzumab was administered IV at a dose of 20 mg/kg weekly (Days 1, 8, 15 and 22 of 4-week cycle) for the first 2 cycles and bi-weekly (every 2 weeks) (Day 1 and Day 15) thereafter until disease progression or unacceptable toxicity became apparent. Lenalidomide 25 mg was administered PO once daily for the first 3 weeks of each 4-week cycle. The dose of lenalidomide was administered at least 2-4 hours after completion of elotuzumab infusion. On weeks without elotuzumab administration, dexamethasone was administered PO as a single dose of 40 mg. On weeks of elotuzumab infusion, the weekly dose of dexamethasone was administered as a split dose of: 28 mg PO (between 3 to 24 hours prior to the start of the elotuzumab infusion) and 8 mg IV (At least 45 min prior to the start of the elotuzumab infusion).
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

3. Secondary Outcome: Number of Participants With Best Overall Response - Treated Participants
Description: Complete response (CR) and Partial Response (PR) were based on the European Group for Blood and Bone Marrow Transplant (EBMT) Criteria. Very Good Partial response was derived from the International Myeloma Working Group (IMWG) criteria. Participants who had a reduction in M-protein or plasmacytoma but did not meet the EBMT criteria for PR were classified as minimal response (MR). Hematologic, radiologic and/or clinical assessments were done every cycle starting with cycle 2. Each cycle is 4 weeks in length (Day 1, Day 8, Day 15, Day 22). Cycle 2 began on study Day 29. CR=negative immunofixation 6 weeks, <5% plasma cells, no increase in size or number of lytic lesions, complete disappearance of extramedullary plasmacytoma. PR=≥50%reduction in M-protein for 6 weeks, ≥90% reduction of urinary light chain excretion or < 200 mg/24hours for 6 weeks, ≥50% reduction in size of extramedullary plasmacytoma present at baseline, no increase in size or number of lytic lesions.
Time Frame: Cycle 2 (Study Day 29) to last dose (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized (Treated Participants).
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants
  Complete Response | 0 | 1
  Very Good Partial Response | 1 | 2
  Partial Response | 1 | 0
  Minimal Response | 1 | 0

4. Secondary Outcome: Geometric Mean Maximum Observed Serum Elotuzumab Concentration (Cmax) During Cycles 1, 2, and 3
Description: The quantification of elotuzumab in human serum was performed using a validated enzyme-linked immunosorbent assay (ELISA). Cmax was measured in micrograms per milliliter (µg/mL). Samples of serum were obtained at: Cycle 1, Day 1: 0 hour (h), 30 minutes (min) 2 h post dose; Day 8: 0h, 2 h; Day 15: 0h, 30 min; Day 22: 0h, 30min, 2h. Cycle 2, Day 1, 22 0h, 2h. Cycle 3, Day 1: 0h, 30h, 2h; Day 15: 0h.
Time Frame: Days 1, 8, 15 and 22 of cycle 1, Days 1 and 22 of cycle 2, Days 1 and 15 of cycle 3
Population: All participants who received at least one dose of study medication and had adequate Pharmacokinetic (PK) concentration profiles were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
µg/mL
  Cycle 1 Day 1 (n=3,3) | 173 (9) | 376 (14)
  Cycle 1 Day 8 (n=3,3) | 237 (19) | 549 (18)
  Cycle 1 Day 15 (n=3,3) | 297 (10) | 652 (21)
  Cycle 1 Day 22 (n=3,2) | 234 (14) | 724 (45)
  Cycle 2 Day 1 (n=3,3) | 240 (28) | 671 (51)
  Cycle 2 Day 22 (n=3,3) | 270 (32) | 844 (26)
  Cycle 3 Day 1 (n=3,3) | 286 (32) | 972 (32)

5. Secondary Outcome: Geometric Mean Minimum Observed Serum Elotuzumab Concentration (Cmin) During Cycles 1, 2, and 3
Description: The quantification of elotuzumab in human serum was performed using a validated enzyme-linked immunosorbent assay (ELISA). Cmin was measured in micrograms per milliliter (µg/mL). Samples of serum were obtained at: Cycle 1, Day 1: 0 hour (h), 30 minutes (min) 2 h post dose; Day 8: 0h, 2 h; Day 15: 0h, 30 min; Day 22: 0h, 30min, 2h. Cycle 2, Day 1, 22 0h, 2h. Cycle 3, Day 1: 0h, 30h, 2h; Day 15: 0h.
Time Frame: Days 8, 15 and 22 of cycle 1, Days 1 and 22 of cycle 2, Days 1 and 15 of cycle 3
Population: All participants who received at least one dose of study medication and had adequate PK concentration profiles were summarized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
µg/mL
  Cycle 1 Day 8 (n=3,3) | 59.1 (28) | 165 (20)
  Cycle 1 Day 15 (n=3,3) | 97.0 (12) | 252 (30)
  Cycle 1 Day 22 (n=3,2) | 24.6 (87) | 280 (62)
  Cycle 2 Day 1 (n=3,2) | 25.8 (95) | 389 (64)
  Cycle 2 Day 22 (n=3,3) | 57.8 (82) | 547 (41)
  Cycle 3 Day 1 (n=3,3) | 77.2 (78) | 579 (46)
  Cycle 3 Day 15 (n=3,3) | 59.4 (78) | 466 (38)

6. Primary Outcome: Number of Participants With Worst Toxicity Grade Hematology Laboratory Tests
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 was used to measure toxicity scale. Lower Limits of Normal (LLN). Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL. Lymphocytes (absolute) Gr 1: <1.5 to 0.8 *10^3 c/µL, Gr 2 <0.8 to 0.5 *10^3 c/µL, Gr 3: <0.5 to 0.2 *10^3 c/µL, Gr 4: <0.2*10^3 c/µL. Neutrophils (absolute): Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Leukocytes Gr 1:<LLN to 3.0 *10^3 c/µL, Gr 2; <3.0 to 2.0 *10^3 c/µL, Gr 3: <2.0 to 1.0 *10^3 c/µL, Gr 4: <1.0 *10^3 c/µL.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants
  Hemoglobin Any Grade | 3 | 3
  Hemoglobin Grade 3-4 | 0 | 1
  Lymphocytes Any Grade | 3 | 3
  Lymphocytes Grade 3-4 | 3 | 3
  Neutrophils Any Grade | 3 | 3
  Neutrophils Grade 3-4 | 2 | 3
  Platelet Count Any Grade | 3 | 2
  Platelet Count Grade 3-4 | 1 | 0
  Leukocytes Any Grade | 3 | 3
  Leukocytes Grade 3-4 | 2 | 1

7. Primary Outcome: Number of Participants With Worst Toxicity Grade Renal and Liver Function Laboratory Tests
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 was used to measure toxicity scale. Lower Limits of Normal (LLN). Upper Limits of Normal (ULN). Alanine transaminase (ALT); Aspartate aminotransferase (AST); Alkaline phosphatase (ALP). ALT Grade (Gr)1:>1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. AST Gr 1: >1.0 to 2.5*ULN; Gr 2: >2.5 to 5.0*ULN; Gr 3: >5.0 to 20.0*ULN; Gr 4: >20.0*ULN. Total bilirubin Gr 1: >1.0 to 1.5*ULN; Gr 2: >1.5 to 3.0*ULN; Gr 3: >3.0 to 10..0*ULN; Gr 4: >10.0.0*ULN. ALP (U/L) Gr1:>1.0 to 2.5*ULN, Gr2:>2.5 to 5.0*ULN, Gr3:>5.0 to 20.0*ULN, Gr4:>20.0*ULN. Albumin (low) Gr 1:<LLN to 3 grams per deciliter (g/dL); Gr 2: <3.0 - 2.0 g/L; Gr 3: < 2 g/dL. Creatinine Gr 1: >1 - 1.5*baseline (BL)to >ULN - 1.5*ULN; Gr 2: >1.5 - 3.0*BL to > 1.5 - 3.0*ULN; Gr 3: >3.0*BL to > 3.0 - 6.0*ULN; Gr 4: >6.0*ULN.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants
  Albumin Any Grade | 3 | 3
  Albumin Grade 3-4 | 0 | 0
  ALP Any Grade | 1 | 2
  ALP Grade 3-4 | 0 | 0
  ALT Any Grade | 2 | 2
  ALT Grade 3-4 | 1 | 1
  AST Any Grade | 1 | 2
  AST Grade 3-4 | 1 | 1
  Creatinine Any Grade | 0 | 2
  Creatinine Grade 3-4 | 0 | 0
  Bilirubin Total Any Grade | 1 | 0
  Bilirubin Total Grade 3-4 | 0 | 0

8. Primary Outcome: Number of Participants With Worst Toxicity Grade Chemistry Laboratory Tests
Description: NCI CTCAE, version 3.0 was used to measure toxicity scale. Sodium high (H) Gr 1:>ULN - 150; Gr 2: >150 - 155; Gr 3: >155 - 160; Gr 4: >160 mmol/L; Sodium low(L) Gr 1:<LLN - 130; Gr 3: <130 - 120; Gr 4: <120 mmol/L. Potassium (H) Gr 1: >ULN - 5.5; Gr 2: >5.5 - 6.0; Gr 3: > 6.0 - 7.0; Gr 4: >7.0 mmol/L; Potassium (L) Gr 1 - Gr 2: <LLN - 3.0; Gr 3: < 3.0 - 2.5; Gr 4: <2.5 mmol/L.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants
  Potassium High, Any Grade | 0 | 2
  Potassium High, Grade 3-4 | 0 | 0
  Potassium Low, Any Grade | 3 | 2
  Potassium Low, Grade 3-4 | 0 | 1
  Sodium High, Any Grade | 1 | 2
  Sodium High, Grade 3-4 | 0 | 0
  Sodium Low, Any Grade | 2 | 3
  Sodium Low, Grade 3-4 | 0 | 0

9. Secondary Outcome: Number of Participants Positive for Anti-Elotuzumab Anti-drug Antibodies - Treated Participants
Description: The detection of anti-elotuzumab anti-drug antibodies (ADAs) in human serum was performed using a validated bridging electrochemiluminescence immunoassay (ECLA) on the Meso Scale Discovery (MSD) platform. Sample collection was performed prior to administration of elotuzumab at Day 1 of each cycle.
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Population: All participants who received at least one dose of study medication were summarized.
Measure: Number; unit: participants
Arm/Group | Elotuzumab 10 mg/kg | Elotuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3
participants | 3 | 0

ADVERSE EVENTS:
Time Frame: First dose (Day 1) to last dose plus 60 days (assessed up to January 2017, approximately 71 months)
Arm/Group | BMS 10mg/kg + Ld | BMS 20mg/kg + Ld
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 10mg/kg + Ld (N=3) | BMS 20mg/kg + Ld (N=3)
Cataract (Eye disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS 10mg/kg + Ld (N=3) | BMS 20mg/kg + Ld (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 3
Lymphopenia (Blood and lymphatic system disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Dental caries (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gingival erosion (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral fungal infection (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 1
Electrocardiogram qt prolonged (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subepidermal (Skin and subcutaneous tissue disorders) | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Flushing (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.